CLINICAL TRIAL: NCT05751083
Title: Effects of Brisk Walk With Low Intensity Aerobic Exercises on Flexibility, Balance, Muscle Endurance and Life Satisfaction in Elderly
Brief Title: Effects of Brisk Walk With Low Intensity in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AQIB SAGHEER REC-014111
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Healthy Aging
Keywords: aerobic exercises; flexibility; balance; endurance; satisfaction; elderly
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- brisk walk+ low intensity aerobic exercises group (Experimental): this group will perform the following exercises Brisk Walking Protocol
  The brisk walking protocol will consist of :
  1. 10 min of warm-up period with flexibility exercises of the knees, hips and back
  2. 30 min of walking
  3. 5 min of cool down.
  General flexibility Exercises Protocol Chair Sitting exercise Standing Balance Exercises
  Interventions: Other: brisk walk+ low intensity aerobic exercises
- brisk walk group (Active Comparator): this group will perform the following exercises Brisk Walking Protocol
  The brisk walking protocol will consist of :
  1. 10 min: warming up of the knees, hips and back by flexibility exercises
  2. 30 min of walking
  3. 5 min of cool down.
  Interventions: Other: Brisk walk

INTERVENTIONS:
Other: brisk walk+ low intensity aerobic exercises — Brisk Walking Protocol General flexibility Exercises Protocol Chair Sitting
  1. Extending leg up then down
  2. Raising up then down on toes later heels
  3. Marching in place
  4. Bringing leg to sideway then back towards middle
  5. Bringing leg towards chair then forward
  6. Bend arms up towards shoulders then back down again.
  7. Pushing arms away from chest then back
  8. Pushing arm up from shoulders then back down
  9. Raising shoulders towards ears then back down
  10. Rolling shoulders forward and backward
  11. Raising arm at shoulder levels and extend forearm upward towards ceiling then back down
  12. Bringing elbows inwards and outwards from chest Standing Balance Exercises
  Arms: brisk walk+ low intensity aerobic exercises group
Other: Brisk walk — Brisk Walking Protocol
  The brisk walking protocol will consist of :
  1. 10 min: warming up of the knees, hips and back by flexibility exercises
  2. 30 min of walking
  3. 5 min of cool down.
  Arms: brisk walk group

SUMMARY:
The goal of this clinical trial is to compare the effects of brisk walk with low intensity aerobic exercises on flexibility balance muscle endurance and life satisfaction in healthy elderly population. The main question it aims to answer is:

• Is brisk walk with low intensity aerobic exercises will improve flexibility, balance, muscle endurance and life satisfaction in healthy elderly population.

Participants will be divided into Group A and Group B. Group A will perform brisk walk with low intensity exercises while group B will perform only brisk walk.

DETAILED DESCRIPTION:
According to world population ageing, the worldwide populace aged equal to and greater than 60 years counted 9.62 × 108 as of 2017. It is contemplated to twofold by 2050 and is estimated to attain 2.1 billion. Regionally, in the emerging countries, there is rapid increase in the percentage at which the inhabitants are ageing, with Asia where a substantial number of individuals fall in the age category of 60 years and above. In Pakistan the longevity in previous 50 years has raised by thirty years, and it is expected to stretch to 72 years by 2023. Pakistan, being the world's sixth most populace, as of now has greater than 8 million elderly individuals and this count is likely to get to 27 million by 2050. Generally, there is declination of physical activity and wellbeing as one ages; nevertheless, evaluation of the effect of sedentary lifestyle on population health often neglect to especially target elderly. Literature recommends that the age specific reduction in functional capacity, quality of life, and expanded risk of morbidity, handicap, and mortality might be counterbalanced or postponed by the acquisition of more physical activity. Nonetheless, physical inactivity has become almost omnipresent, with an expected 31% of the total populace not gathering suggested physical activity levels.

Evolving evidence showed a weekly performance of moderate to vigorous physical activities for 75 minutes per week has been related with a decrease in all-cause mortality by 22% in elderly aged ≥60 years. The WHO has recommended that taking part in moderate-to-vigorous physical activity for 150 minutes out of every week, with every session enduring at the very least 10 minutes, will prompt good health. It is sufficiently accepted that the musculoskeletal framework contributes a significant part in the falling mechanics. The functional outcome of the musculoskeletal framework is decreased in the older population. Predominantly, overall motor function of the lower limbs reduces, and muscle strength declines There is insufficient data on the effect of low intensity exercise on flexibility, balance, muscle endurance and life satisfaction, particularly in healthy older males. Moreover, there is no study conducted up until now, on the combined effect of brisk walking and low aerobic exercises on varied variables in the elderly. This study will contribute by examining the effectiveness of brisk walking along with low intensity aerobic exercises on flexibility, balance, muscle endurance and life satisfaction in the older male population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60
* Gender: Male
* Healthy adults
* Participants who have no medical condition according to the pre-screening tool PAR-Q+.

Exclusion Criteria:

* Diagnosed cases of 3rd or 4th stage osteoporosis
* Obese (BMI > 30)
* Systemic disorders, Trauma, Disability
* Cancer, Musculoskeletal disorders

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The Physical Activity Readiness Questionnaire for Everyone PAR-Q+ | Twelve weeks
  It screens for any risks while performing moderate physical activity and reviews family history and severity of the disease. The reliability of this questionnaire was high (r = 0.99)
Modified Wells Bench Test | Twelve weeks
  It is used to measure the flexibility of the lower back and hamstrings. The participant is sitting on the ground with legs extended forward and supported against the box. The individual is instructed to reach forward and perform flexion of the trunk, obtaining a score in centimeter. It has good intraclass test-retest reliability R = .92 and moderate-to-good relation with the criterion measure r = .76 for male elderly
6 min walk test | Twelve weeks
  The 6 Minute Walk Test is a test used to measure aerobic capacity as well as endurance. The covered distance of 6 minutes is used as the outcome to correlate changes in performance capacity. It has excellent test-retest reliability (ICC =0.95)
The Mini-BESTest | Twelve weeks
  It was developed in 2010 by Franchignoni et al. This clinical balance assessment tool is a shortened version of Balance Evaluation Systems (BESTest). This scale assesses dynamic balance , a unidimentional construct and includes 14 items addressing 4 sections; 1) Anticipatory postural adjustment 2) Reactive postural control 3)Sensory orientation 4) Dynamic gait. It has excellent test-retest reliability ICC =0.96 and validity r=0.72 (CI 0.61-0.81)
Satisfaction with life scale | Twelve weeks
  It is a brief 5-item tool devised to evaluate participant's perceived satisfaction with life. The SWLS is a 7-point Likert style response scale. It has adequate validity r=(0.81)

CONTACTS AND LOCATIONS:
Overall Officials: Aadil Omer, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Shahid international gym rawalpindi, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No